CLINICAL TRIAL: NCT06616116
Title: Development and Verification of Effectiveness of Biofeedback Contents for Stress Management Using Real-time Bio-signal Monitoring Device
Brief Title: Stress Management with Real-time Bio-signal Biofeedback
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyunju Lee, Principal Investigator, MD., PhD, Assistant Professor of Clinical Psychiatry, Department of Psychiatry, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RS-2023-00279070
Record Dates: First submitted 2024-09-06; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Bipolar Disorder (BD); Major Depressive Diorder
Keywords: biosignal; neurofeedback; mindfulness; bipolar disorder; major depressive disorder
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder, Major | interventions — Biofeedback, Psychology; Neurofeedback; Real-Time Polymerase Chain Reaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness with biosignal feedback (Experimental): Biosignal Monitoring (EEG and HRV) with Real-time neurofeedback during Mindfulness
  Interventions: Device: Biosignal feedback
- Mindfulness without biosignal feedback (Sham Comparator): Biosignal Monitoring (EEG and HRV) without Real-time neurofeedback during Mindfulness
  Interventions: Device: Sham Comparator

INTERVENTIONS:
Device: Biosignal feedback — 1. Real-time neurofeedback guided mindfulness
     : Unlike standard mindfulness therapies, this intervention integrates real-time monitoring of brainwave activity (EEG). Participants in the experimental group receive immediate auditory feedback during their mindfulness sessions, which helps guide their practice and enhance engagement.
  2. Tailored progress report In addition to real-time feedback, participants in the Mindfulness with biosignal feedback group receive detailed reports of their biosignal data (EEG and HRV) before, during, and after each session. These reports allow for deeper self-reflection and personalized adjustments to their mindfulness practice, which is not commonly provided in other mindfulness programs.
  Other Names: biofeedback; neurofeedback; real-time
  Arms: Mindfulness with biosignal feedback
Device: Sham Comparator — Biosignal Monitoring (EEG and HRV) during Mindfulness without real-time feedback
  Other Names: Biosignal monitoring only
  Arms: Mindfulness without biosignal feedback

SUMMARY:
The goal of this clinical trial is to learn if the real-time bio-signal monitoring device (Neuronicle FX2 device), combined with mindfulness-based cognitive therapy (MBCT), helps manage stress and improves symptoms of mood disorders, such as depression and anxiety. The main questions this study aims to answer are:

* Does real-time bio-signal feedback mindfulness using the Neuronicle FX2 reduce perceived stress in participants with mood disorders?
* Does it lead to improvements in depressive and anxiety symptoms?

Researchers will compare participants receiving real-time biofeedback with the Neuronicle FX2 to those receiving no feedback during mindfulness sessions to see if the device enhances the effectiveness of stress management and symptom improvement.

Participants will:

* Undergo mindfulness-based cognitive therapy (MBCT) once a week for 8 weeks.
* Half of the participants will receive real-time biofeedback using the Neuronicle FX2 device during mindfulness sessions, while the other half will not be provided biofeedback.
* Visit the clinic every week for their mindfulness sessions and assessments.
* Wear the Neuronicle FX2 device during mindfulness exercises, which will measure brainwave activity (EEG) and heart rate variability (HRV).
* Participate in assessments before, during, and after the program (8wks, 16wks) to evaluate their stress, depression, and anxiety levels.

DETAILED DESCRIPTION:
This clinical trial aims to evaluate the effectiveness of biosignal guided Mindfulness-based Cognitive Therapy (MBCT) in managing stress and improving mood disorder symptoms in participants aged 15 to 60, who are diagnosed with mood disorders such as major depressive disorder and bipolar disorder.

Participants will be randomly assigned to one of two groups:

1. Biosignal-guided group: Participants will receive real-time biofeedback during mindfulness exercises. This feedback, derived from biosignals like brainwave activity (EEG), will help guide their mindfulness practice. In addition, participants in this group will receive a report summarizing their EEG and HRV data before, during, and after each mindfulness session to track their progress and provide insights into their physiological responses.
2. Standard group: Participants will engage in the same mindfulness exercises, but without receiving real-time feedback. Their biosignals will still be monitored for comparative purposes.

The primary goal of this study is to determine whether real-time biosignal feedback can enhance the effectiveness of mindfulness in reducing perceived stress. Secondary outcomes include changes in depressive and anxiety symptoms. These will be assessed using validated measures like the Korean Perceived Stress Scale (K-PSS), Hamilton Depression Rating Scale (HAM-D), and others.

The trial will run for 8 weeks, with weekly mindfulness sessions. Follow-up assessments will be conducted at 8 and 16 weeks post-intervention to evaluate the long-term effects of the therapy.

This research seeks to contribute to the development of personalized stress management interventions by using biosignal-guided mindfulness as a tool to improve treatment adherence and effectiveness in managing mood disorders.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 15 to 59 years.
* Patients diagnosed with mood disorders (e.g., bipolar disorder, major depressive disorder) through screening and clinician interviews, according to DSM-5.
* Patients with accompanying anxiety symptoms.
* Patients with stress symptoms (Perceived Stress Scale score ≥ 10)
* Individuals able to independently complete questionnaires and communicate in Korean.
* Individuals who voluntarily agree to participate in weekly treatment sessions.

Exclusion Criteria:

* Patients diagnosed with major psychiatric disorders other than mood disorders (e.g., schizophrenia, substance use disorders including alcohol, obsessive-compulsive disorder).
* Patients diagnosed with bipolar disorder who are currently experiencing acute psychotic symptoms or are in a manic state.
* Individuals with acute suicidal ideation.
* Individuals with co-occurring personality disorders (e.g., borderline personality disorder, antisocial personality disorder, narcissistic personality disorder).
* Individuals who have participated in mindfulness-based cognitive therapy within the last 3 months.
* Individuals currently receiving other non-pharmacological treatments (e.g., cognitive-behavioral therapy, psychoanalysis).
* Individuals with neurological damage or conditions that may cause brain injury (e.g., seizure disorder, cerebrovascular or neoplastic lesion, neurodegenerative disorder, significant head trauma with loss of consciousness lasting more than 5 minutes).
* Individuals diagnosed with cardiovascular diseases (e.g., hypertension, coronary artery disease, arrhythmia).
* Individuals with hearing impairment or tinnitus.
* Individuals with impaired ability to understand the study's purpose or make decisions about participation (e.g., IQ < 70, dementia).
* Individuals with medical, psychological, social, or legal issues that would interfere with continued participation in the program.

Ages: 15 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline Korean Perceived Stress Scale (K-PSS) score at 8wks, and 16 wks | Baseline (pre-treatment), immediately after the 8-week intervention, and at 2-month follow-up.
  The full name: Perceived Stress Scale - 10 item form 14-item scale developed by Cohen et al. (1983) that emphasizes subjective perception of stress. Measures the degree of perceived unforeseeable, uncontrollable, and overwhelming experience of stress in the past month. Although the 14-item PSS tend to exhibit good reliability, four of the items tend to perform poorly when evaluated using exploratory factor analysis (Cohen et al., 1988). As a result, the PSS is commonly implemented using the 10-item form. The questions are rated on 5-point Likert scale; 0 (never), 1 (almost never), 2 (sometimes), 3 (fairly often), 4 (very often). Higher scores represent worse outcomes. The scores of each scale sum into the total score. Thus the total score ranges from 0 to 40.

SECONDARY OUTCOMES:
Change from baseline Inventory of Depressive Symptomatology (IDS-SR) score | Baseline, immediately after the 8-week intervention, and at 2-month follow-up.
  The Inventory of Depressive Symptomatology-Self Report (IDS-SR) is a self-report questionnaire used to assess the severity of depressive symptoms. It was developed to provide a comprehensive evaluation of various dimensions of depression, including mood, cognition, behavior, and physical symptoms.
  IDS-SR16 version is used for this study: A shorter, 16-item version focusing on core depressive symptoms.
Change from baseline Hamilton depression rating scale (HAM-D) score | Baseline, immediately after the 8-week intervention, and at 2-month follow-up.
  The Hamilton Depression Rating Scale (HAM-D) is a 17-item assessment tool used by interviewers to evaluate the severity of depressive symptoms. According to the reliability and validation study of the Korean version, the internal consistency reliability was 0.76. The total score ranges from 0 to 52, with higher scores indicating more severe depression.
Change from baseline Hamilton anxiety rating scale (HAM-A) score | Baseline, immediately after the 8-week intervention, and at 2-month follow-up.
  The Hamilton Anxiety Rating Scale (HAM-A) is an interviewer-administered assessment tool used to evaluate the severity of anxiety symptoms over the past 7 days. It consists of 14 items and includes both psychological and physical anxiety symptoms. Each item is rated on a scale from 0 to 4, with the total score ranging from 0 to 56, where higher scores indicate more severe anxiety.
Change from baseline Anxiety Sensitivity Index (ASI)score | Baseline, immediately after the 8-week intervention, and at 2-month follow-up.
  The ASI consists of 16 items, each rated on a scale from 0 (very little) to 4 (very much), where respondents indicate how much they agree with statements about their anxiety-related concerns. The total score ranges from 0 to 64, with higher scores reflecting greater anxiety sensitivity.
Change from baseline Generalized Anxiety Disorder-7 (GAD-7) score | Baseline, immediately after the 8-week intervention, and at 2-month follow-up.
  The Generalized Anxiety Disorder-7 (GAD-7) is a widely used self-report questionnaire designed to assess the severity of generalized anxiety disorder (GAD) symptoms. It is brief, consisting of 7 items that focus on key symptoms of anxiety experienced over the past two weeks. Each item in the GAD-7 is scored on a 4-point scale, based on how often the respondent has experienced symptoms. The total score is the sum of the seven items, giving a range from 0 to 21, with higher scores indicating more severe anxiety.
Change from baseline Young Mania Rating Scale (YMRS) score | Baseline, immediately after the 8-week intervention, and at 2-month follow-up.
  The Young Mania Rating Scale (YMRS) is a clinician-administered tool used to assess the severity of manic symptoms in individuals with bipolar disorder. It is one of the most widely used rating scales for mania and is particularly useful in both clinical and research settings to evaluate treatment effects or monitor symptom changes over time. The YMRS consists of 11 items, each focusing on different aspects of mania, such as mood, behavior, and cognitive functioning. These items are rated by the clinician based on the individual's behavior and self-report of symptoms over the past 48 hours.
  The scoring is based on a 0 to 4 scale for most items, but four items (irritability, speech, thought content, and disruptive/aggressive behavior) are scored on a 0 to 8 scale, to give more weight to these important aspects of mania.
Change from baseline Beck Scale for Suicide Ideation(SSI-Beck) score | Baseline, immediately after the 8-week intervention, and at 2-month follow-up.
  The Scale for Suicide Ideation (SSI), often referred to as the Beck Scale for Suicide Ideation (SSI-Beck), is a clinical tool used to assess the intensity, frequency, and characteristics of suicidal thoughts in individuals. Developed by Aaron T. Beck and colleagues, it is designed to measure the severity of both active and passive suicidal ideation.
  The SSI-Beck consists of 19 items, each assessing different aspects of suicidal ideation. Each item is rated on a 3-point scale (from 0 to 2), with higher scores indicating greater severity of suicidal thoughts or intent. The total score ranges from 0 to 38, with higher scores suggesting a higher risk of suicide.
Change from baseline Patient Health Questionnaire-15 (PHQ-15) score | Baseline, immediately after the 8-week intervention, and at 2-month follow-up.
  The Patient Health Questionnaire-15 (PHQ-15) is a self-report questionnaire designed to assess the severity of somatic symptoms, particularly in patients who may have somatization disorders or other medically unexplained physical symptoms. It is part of the broader PHQ suite of tools used for assessing various aspects of mental health.
  The PHQ-15 consists of 15 items, each related to common physical symptoms that can be associated with psychological distress. Patients rate how much they have been bothered by these symptoms over the past four weeks on a 3-point scale. The total score is calculated by summing the responses, with a range from 0 to 30. Higher scores indicate a greater severity of somatic symptoms.
Change from baseline World Health Organization Quality of Life-BREF (WHOQOL-BREF) score | Baseline, immediately after the 8-week intervention, and at 2-month follow-up.
  The World Health Organization Quality of Life-BREF (WHOQOL-BREF) is a self-report questionnaire designed to assess an individual's quality of life across various domains. It is a shorter version of the original WHOQOL-100 and is used in both clinical settings and research to evaluate general well-being and life satisfaction in relation to health. The WHOQOL-BREF contains 26 items, which measure quality of life in four main domains: Physical health (7 items), Psychological Health (6 items), Social relationships (3 items), and Environment (8 items). Each item is rated on a 5-point Likert scale, where respondents rate how much they agree with statements or how satisfied they are with certain aspects of their life. Scores are then transformed to reflect a scale of 0 to 100, with higher scores indicating better quality of life.
Change from baseline Five-Factor Mindfulness Questionnaire (FFMQ-Short Form) score | Baseline, immediately after the 8-week intervention, and at 2-month follow-up.
  The Five-Factor Mindfulness Questionnaire-Short Form (FFMQ-SF) is a condensed version of the original FFMQ, designed to assess the extent to which individuals engage in mindful behavior. The full FFMQ was based on five key aspects of mindfulness derived from multiple sources of mindfulness measurement, and the short form provides a more concise tool for measuring mindfulness in research and clinical settings. The FFMQ-SF consists of 24 items, divided into five subscales representing different facets of mindfulness. Each item is rated on a 5-point Likert scale. The total score and subscale scores are calculated by summing the individual items. Higher scores indicate a higher level of mindfulness.
Change from baseline Cognitive and Affective Mindfulness Scale-Revised (CAMS-R) score | Baseline, immediately after the 8-week intervention, and at 2-month follow-up.
  The Cognitive and Affective Mindfulness Scale-Revised (CAMS-R) is a self-report questionnaire that assesses mindfulness, focusing on the individual's ability to regulate attention and maintain awareness of the present moment. The Korean version, K-CAMS-R, is an adaptation of the original CAMS-R to ensure cultural relevance and language consistency for Korean-speaking populations.
  The K-CAMS-R consists of 10 items that measure key aspects of mindfulness. Each item is rated on a 4-point Likert scale, indicating the degree to which the statement applies to the respondent. The total score is the sum of the item scores, with higher scores reflecting greater mindfulness.
Heart Rate Variability (HRV) | Baseline, immediately after the 8-week intervention, and at 2-month follow-up.
  HRV is recorded with a device (neuroNicle FX2, Laxtha) which include EEG and HRV recording system. HRV is calculated from pulse rate signal recorded at earlobe.
Quantitative electroencephalography (QEEG) | Baseline, immediately after the 8-week intervention, and at 2-month follow-up.
  EEG is recorded with a device (neuroNicle FX2, Laxtha) which include EEG and HRV recording system. EEG signal is acquired at the prefrontal area, two channels (FP1, FP2) on forehead.
  Power spectrum analysis of the EEG data will be performed using Fourier analysis. And absolute power, relative power, of each frequency band, symmetry are included.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea